CLINICAL TRIAL: NCT06244693
Title: Description and Analysis of Congestion During Hospitalization for Acute Decompensated Heart Failure
Brief Title: SUbCONgestion in Heart Failure Registry
Acronym: SUCONIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2024
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure; Congestion
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Analytical measurements from blood samples for biomarkers, not DNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to learn about the decongestion process in heart failure patients. The main question it aims to answer is: What is the behavior of congestion during hospitalization in adult patients with acute heart failure (AHF)? Participants will be evaluated in the decongestion process through clinical, analytical, and ultrasonographic variables, and they will be followed up for one year to assess mortality and rehospitalization rates in this population.

DETAILED DESCRIPTION:
Heart failure (HF) is a syndrome characterized by the presence of dyspnea, lower extremity edema, orthopnea, jugular venous distention, and pulmonary crackles, among others, secondary to elevated ventricular filling pressures. It is the leading cause of hospitalization in medical services in Chile and worldwide, with the majority of patients being elderly. Decompensation of HF is explained in most cases by fluid overload (congestion) and can be studied through biomarkers, clinical signs, radiographic, and ultrasonographic findings. The Chilean demographic transition makes it necessary to optimize the multiparametric and protocolized management of hospitalized patients.

General Objective: To evaluate and describe the decongestion process, including residual congestion, during hospitalization for heart failure at the Clinical Hospital of the University of Chile (HCUCh).

A prospective observational cohort study will be conducted with all patients hospitalized for heart failure at HCUCh. Clinical, analytical, and ultrasonographic variables, especially those related to congestion assessment, will be recorded. Enrollment will last for one year from institutional authorization, and telephone follow-up will be conducted for one year post-discharge, extendable up to five year.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with decompensated heart failure in the emergency department or cardiology outpatient clinic at the Clinical Hospital of the University of Chile (HCUCh).
* Profile of warm-wet and cold-wet type heart failure.
* Spontaneous ventilation with or without non-invasive mechanical support.
* Desire for participation validated through informed consent.

Exclusion Criteria:

* Dry-type heart failure profile (warm and cold)
* Diagnostics that mimics heart failure (valvular heart disease, cardiomyopathies, and others diagnostic different from heart failure).
* Septic, distributive, or obstructive shock
* Polytraumatized
* Severe burns
* Invasive mechanical ventilation
* Permanent renal replacement therapy
* Severe dependence
* Presence of terminal illness with a prognosis of survival less than one year
* Presence of traumatic conditions that prevent the use of thoracic ultrasound, such as a flail chest or moderate to severe burn on the left hemithorax.
* Lack of a support network or contact.
* Cardiorespiratory arrest
* Refusal to participate as indicated in the informed consent.
* Presence of psychological or intellectual disability that prevents expressing the will to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure aged 18 years or above that are admitted in emergency room or outpatient clinic for acute decompensation of new or known heart failure, excluding diagnostics that mimics heart failure. Everyone has to be discharge from Hospital Clínico Universidad de Chile.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization | One year from discharge
  Readmission to hospital for cardiac cause
All cause mortality | One year after discharge
  Death from any cause

SECONDARY OUTCOMES:
Cardiac death | One year after discharge
  Death form cardiac cause

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Parra, MD,PhD, Principal Investigator — Departamento Cardiovascular - Hospital Clínico Universidad de Chile
Locations (1):
- Departamento Cardiovascular - Hospital Clínico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
Use data for compare with other populations in other studies.

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Roger VL. Epidemiology of heart failure. Circ Res. 2013 Aug 30;113(6):646-59. doi: 10.1161/CIRCRESAHA.113.300268. PMID 23989710
- [Background] Castro P, Vukasovic JL, Garces E, Sepulveda L, Ferrada M, Alvarado S; Insuficiencia Cardiaca: Registro y Organizacion. [Cardiac failure in Chilean hospitals: results of the National Registry of Heart Failure, ICARO]. Rev Med Chil. 2004 Jun;132(6):655-62. doi: 10.4067/s0034-98872004000600001. Spanish. PMID 15332366
- [Background] Diaz-Toro F, Nazzal N C, Verdejo P H. [Incidence and hospital mortality due to heart failure. Are there any differences by sex?]. Rev Med Chil. 2017 Jun;145(6):703-709. doi: 10.4067/s0034-98872017000600703. No abstract available. Spanish. PMID 29171617
- [Background] Selvaraj S, Claggett B, Pozzi A, McMurray JJV, Jhund PS, Packer M, Desai AS, Lewis EF, Vaduganathan M, Lefkowitz MP, Rouleau JL, Shi VC, Zile MR, Swedberg K, Solomon SD. Prognostic Implications of Congestion on Physical Examination Among Contemporary Patients With Heart Failure and Reduced Ejection Fraction: PARADIGM-HF. Circulation. 2019 Oct 22;140(17):1369-1379. doi: 10.1161/CIRCULATIONAHA.119.039920. Epub 2019 Sep 12. PMID 31510768
- [Background] Pan D, Pellicori P, Dobbs K, Bulemfu J, Sokoreli I, Urbinati A, Brown O, Sze S, Rigby AS, Kazmi S, Riistama JM, Cleland JGF, Clark AL. Prognostic value of the chest X-ray in patients hospitalised for heart failure. Clin Res Cardiol. 2021 Nov;110(11):1743-1756. doi: 10.1007/s00392-021-01836-9. Epub 2021 Mar 22. PMID 33754159
- [Background] Ambrosy AP, Cerbin LP, Armstrong PW, Butler J, Coles A, DeVore AD, Dunlap ME, Ezekowitz JA, Felker GM, Fudim M, Greene SJ, Hernandez AF, O'Connor CM, Schulte P, Starling RC, Teerlink JR, Voors AA, Mentz RJ. Body Weight Change During and After Hospitalization for Acute Heart Failure: Patient Characteristics, Markers of Congestion, and Outcomes: Findings From the ASCEND-HF Trial. JACC Heart Fail. 2017 Jan;5(1):1-13. doi: 10.1016/j.jchf.2016.09.012. PMID 28034373
- [Background] Wettersten N. Biomarkers in Acute Heart Failure: Diagnosis, Prognosis, and Treatment. Int J Heart Fail. 2021 Feb 15;3(2):81-105. doi: 10.36628/ijhf.2020.0036. eCollection 2021 Apr. PMID 36262882
- [Background] Fonarow GC, Abraham WT, Albert NM, Gattis WA, Gheorghiade M, Greenberg B, O'Connor CM, Yancy CW, Young J. Organized Program to Initiate Lifesaving Treatment in Hospitalized Patients with Heart Failure (OPTIMIZE-HF): rationale and design. Am Heart J. 2004 Jul;148(1):43-51. doi: 10.1016/j.ahj.2004.03.004. PMID 15215791
- [Background] Ibrahim NE, Januzzi JL Jr. Beyond Natriuretic Peptides for Diagnosis and Management of Heart Failure. Clin Chem. 2017 Jan;63(1):211-222. doi: 10.1373/clinchem.2016.259564. Epub 2016 Oct 10. PMID 28062619
- [Background] Kumric M, Kurir TT, Bozic J, Glavas D, Saric T, Marcelius B, D'Amario D, Borovac JA. Carbohydrate Antigen 125: A Biomarker at the Crossroads of Congestion and Inflammation in Heart Failure. Card Fail Rev. 2021 Jun 12;7:e19. doi: 10.15420/cfr.2021.22. eCollection 2021 Mar. PMID 34950509
- [Background] D'Aloia A, Faggiano P, Aurigemma G, Bontempi L, Ruggeri G, Metra M, Nodari S, Dei Cas L. Serum levels of carbohydrate antigen 125 in patients with chronic heart failure: relation to clinical severity, hemodynamic and Doppler echocardiographic abnormalities, and short-term prognosis. J Am Coll Cardiol. 2003 May 21;41(10):1805-11. doi: 10.1016/s0735-1097(03)00311-5. PMID 12767668
- [Background] Nunez J, Llacer P, Bertomeu-Gonzalez V, Bosch MJ, Merlos P, Garcia-Blas S, Montagud V, Bodi V, Bertomeu-Martinez V, Pedrosa V, Mendizabal A, Cordero A, Gallego J, Palau P, Minana G, Santas E, Morell S, Llacer A, Chorro FJ, Sanchis J, Facila L; CHANCE-HF Investigators. Carbohydrate Antigen-125-Guided Therapy in Acute Heart Failure: CHANCE-HF: A Randomized Study. JACC Heart Fail. 2016 Nov;4(11):833-843. doi: 10.1016/j.jchf.2016.06.007. Epub 2016 Aug 10. PMID 27522630
- [Background] Nunez J, Minana G, Gonzalez M, Garcia-Ramon R, Sanchis J, Bodi V, Nunez E, Chorro FJ, Llacer A, Miguel A. Antigen carbohydrate 125 in heart failure: not just a surrogate for serosal effusions? Int J Cardiol. 2011 Feb 3;146(3):473-4. doi: 10.1016/j.ijcard.2010.12.027. Epub 2010 Dec 28. No abstract available. PMID 21193243
- [Background] Perez Calvo JI, Rubio Gracia J, Josa Laorden C, Morales Rull JL. Residual congestion and clinical intuition in decompensated heart failure. Rev Clin Esp (Barc). 2019 Aug-Sep;219(6):327-331. doi: 10.1016/j.rce.2019.02.004. Epub 2019 Apr 17. English, Spanish. PMID 31005262
- [Background] Appiani F. [Monitoring decongestion in acute heart failure]. Rev Med Chil. 2022 Apr;150(4):493-504. doi: 10.4067/S0034-98872022000400493. Spanish. PMID 36155759
- [Background] Ambrosy AP, Pang PS, Khan S, Konstam MA, Fonarow GC, Traver B, Maggioni AP, Cook T, Swedberg K, Burnett JC Jr, Grinfeld L, Udelson JE, Zannad F, Gheorghiade M; EVEREST Trial Investigators. Clinical course and predictive value of congestion during hospitalization in patients admitted for worsening signs and symptoms of heart failure with reduced ejection fraction: findings from the EVEREST trial. Eur Heart J. 2013 Mar;34(11):835-43. doi: 10.1093/eurheartj/ehs444. Epub 2013 Jan 4. PMID 23293303
- [Background] Rubio-Gracia J, Demissei BG, Ter Maaten JM, Cleland JG, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Davison BA, Givertz MM, Bloomfield DM, Dittrich H, Damman K, Perez-Calvo JI, Voors AA. Prevalence, predictors and clinical outcome of residual congestion in acute decompensated heart failure. Int J Cardiol. 2018 May 1;258:185-191. doi: 10.1016/j.ijcard.2018.01.067. PMID 29544928
- [Background] Girerd N, Seronde MF, Coiro S, Chouihed T, Bilbault P, Braun F, Kenizou D, Maillier B, Nazeyrollas P, Roul G, Fillieux L, Abraham WT, Januzzi J Jr, Sebbag L, Zannad F, Mebazaa A, Rossignol P; INI-CRCT, Great Network, and the EF-HF Group. Integrative Assessment of Congestion in Heart Failure Throughout the Patient Journey. JACC Heart Fail. 2018 Apr;6(4):273-285. doi: 10.1016/j.jchf.2017.09.023. Epub 2017 Dec 6. PMID 29226815
- [Background] Coiro S, Rossignol P, Ambrosio G, Carluccio E, Alunni G, Murrone A, Tritto I, Zannad F, Girerd N. Prognostic value of residual pulmonary congestion at discharge assessed by lung ultrasound imaging in heart failure. Eur J Heart Fail. 2015 Nov;17(11):1172-81. doi: 10.1002/ejhf.344. Epub 2015 Sep 29. PMID 26417699
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- Available data/document: Individual Participant Data Set: aparral — http://www.redcap.med.uchile.cl — Data registry online system provided by sponsor